CLINICAL TRIAL: NCT03670576
Title: It's Not JUST Idiopathic Pulmonary Fibrosis Study
Acronym: INJUSTIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18014
Record Dates: First submitted 2018-08-06; First posted 2018-09-13 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — Blood Specimen Collection; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (Serum, Plasma) Bronchoscopy Biopsy Samples (Optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: A diagnosis of Fibrotic Lung disease classified in 4 categories, RA-UIP, Asbestosis, Chronic HP and Unclassifiable as agreed by an ILD MDT consensus panel.
  Interventions: Procedure: Optional Bronchoscopy; Other: Quality of Life Questionnaires; Other: Blood Samples for Biomarkers; Other: Home Hand Held Spirometry
- Control: Positive control will be frequency matched to cases of ILD and will be people in secondary care who have an MDT diagnosis of Definite IPF.
  Interventions: Procedure: Optional Bronchoscopy; Other: Quality of Life Questionnaires; Other: Blood Samples for Biomarkers; Other: Home Hand Held Spirometry

INTERVENTIONS:
Procedure: Optional Bronchoscopy — Patients can decide to have an optional bronchoscopy so that samples can be taken for research up to three months from baseline.
Other: Quality of Life Questionnaires — MRC Dyspnoea, SPARC, KBILD and EQ-5D-5L will be administered at baseline, 3 months, 12 months and 24 months,
Other: Blood Samples for Biomarkers — a 40ml research blood sample to be taken at baseline, 3 months, 12 months and 24 months.
Other: Home Hand Held Spirometry — Patients will download an app and are given a small hand held device to record their own spirometry at home. This is blinded for the first three months of the study and then requested a week before and a week after the three follow up points (3m, 12m, 24m)

SUMMARY:
Study of progression of fibrosis in ILD

DETAILED DESCRIPTION:
The overall aims of this study are

* Identify biomarkers and gene expression profiles that determine progressive fibrotic lung disease regardless of aetiology
* To prospectively assess biomarkers which predict progressive fibrosis in patients with fibrosing lung disease of alternate aetiology, including RA-UIP, Asbestosis, Chronic Hypersensitivity Pneumonitis and Unclassifiable fibrotic lung disease
* Investigate genetic associations and epigenetic modifications which affect fibrotic disease severity and progression
* Prospectively evaluate longitudinal disease behaviour in patients with non IPF-fibrotic lung diseases with a view to developing composite clinical end-points for subsequent use in intervention studies in patients

ELIGIBILITY:
Inclusion Criteria

* Male or female aged ≥ 18 years old
* Able and willing to give written informed consent
* Recently diagnosed [defined as diagnostic CT scan or surgical lung biopsy (if applicable) >1st May 2017]
* An MDT diagnosis of fibrotic interstitial lung disease (reticulation, traction +/- honeycombing)

Sub Groups

* Rheumatoid arthritis (rheumatologist diagnosed with anti-CCP antibodies and/or Rheumatoid Factor positive)
* Asbestosis (appropriate occupational history and radiological evidence of asbestos exposure)
* Chronic HP in accordance with consensus criteria (appropriate exposure history, radiological features +/- avian and fungal precipitins)
* Unclassifiable fibrotic lung disease (fibrotic lung disease otherwise unclassifiable despite extensive clinical and radiological examination)
* IPF in accordance with consensus criteria (ATS/ERS/JRS/ALAT guidelines) as controls

Exclusion Criteria:

* Participating in an interventional clinic trial
* Asymptomatic Interstitial Lung Abnormalities (ILA) and normal lung function.
* Change in clinical phenotype from initial radiological diagnosis to screening
* Acute Hypersensitivity Pneumonitis.
* Participants who do not possess a smartphone or have a valid email address (necessary for the home FVC readings)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from ILD and IPF clinics.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2022-11-11 (Estimated); Study Completion 2022-11-11 (Estimated)

PRIMARY OUTCOMES:
Disease Progression | Within 12 months
  Disease progression defined as >10% relative decline in FVC (using either hospital spirometry or home hand held spirometry) or death within 12 months.
Overall Survival | 10 years
  All patients will be tagged at the central NHS registry in order to provide mortality data. For this reason we will need to keep our datasets active for up to 10 years to allow a complete mortality analysis.

SECONDARY OUTCOMES:
Serum and Plasma Biomarkers | Baseline, 3 months, 12 months, 24 months
  SPD, MUC16, CA199, Nordic Neoepitopes

OTHER OUTCOMES:
DLco | Baseline, 3 months, 12 months, 24 months
  Diffusing Capacity of the Lung for Carbon Monoxide
Quality of Life Questionnaires | Baseline, 3 months, 12 months, 24 months.
  Assessment of how the patients well-being may be affected over time by their interstitial lung disease
Domicillary Spirometry | Daily for the first 3 months of study then at 2 week periods around time of planned follow up
  Change in home handheld spirometry values from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (24):
- United Kingdom (24):
  - Queens Hospital Burton, Burton-on-Trent, Derbyshire
  - Kings Mill Hospital, Mansfield, Nottingham
  - Royal United Hospitals Bath NHS Trust, Bath
  - University Hospitals Birmingham, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Southmead Hospital North Bristol, Bristol
  - University Hospitals Coventry and Warwickshire, Coventry
  - Royal Derby Hospital, Derby
  - Royal Devon and Exeter Hospital, Exeter
  - Medway Maritime Hospital, Gillingham
  - Kingston Hospital NHS Foundation Trust, London
  - St Georges Hospital, London
  - North Manchester General Hospital, Manchester
  - Wythenshawe Hospital, Manchester
  - Newcastle Upon Tyne NHS Foundation Trust, Newcastle
  - Northumbria Healthcare NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - South Tyneside District Hospital, South Shields
  - University Hospital of North Tees, Stockton-on-Tees
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - Royal Albert and Edward Infirmary, Wigan
  - New Cross Hospital, Wolverhampton
  - Worcestershire Royal Hospital, Worcester

REFERENCES:
- [Derived] Khan F, Stewart I, Howard L, Barber CM, Borton R, Braybrooke R, Hearson G, Jones S, Maher T, Matthews L, Saini G, Thompson N, Wilson AM, Johnson SR, Jenkins G. Comprehensive characterisation of individuals with fibrotic interstitial lung disease: baseline insights from the INJUSTIS study. BMJ Open Respir Res. 2026 Jan 20;13(1):e003112. doi: 10.1136/bmjresp-2024-003112. PMID 41558800
- [Derived] Khan F, Stewart I, Howard L, McKeever TM, Jones S, Hearson G, Braybrooke R, Edwards C, Jenkins G, Saini G. The Its Not JUST Idiopathic pulmonary fibrosis Study (INJUSTIS): description of the protocol for a multicentre prospective observational cohort study identifying biomarkers of progressive fibrotic lung disease. BMJ Open Respir Res. 2019 Jun 4;6(1):e000439. doi: 10.1136/bmjresp-2019-000439. eCollection 2019. PMID 31258922